CLINICAL TRIAL: NCT00103532
Title: Motivational Enhancement to Promote Health and Reduce Risk in HIV-Infected Youth
Brief Title: Healthy Choices to Promote Health and Reduce Risk in HIV-Infected Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATN 004
Record Dates: First submitted 2005-02-09; First posted 2005-02-10 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: HIV Infection
Keywords: motivational enhancement; health behaviors; risk behaviors
MeSH Terms: conditions — HIV Infections; Health Behavior; Risk-Taking | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Choices - Motivational Enhancement Intervention (Experimental): Motivational enhancement intervention
  Interventions: Behavioral: Healthy Choices - Motivational Enhancement Intervention
- Standard Care (Active Comparator): Standard care/individualized referrals
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Healthy Choices - Motivational Enhancement Intervention — Participants who are randomized to the intervention group will participate in four sessions (over approximately 3 months) of Healthy Choices; a motivational enhancement intervention specifically designed to target multiple risk behaviors in HIV+ youth. Participants will receive individualized referrals at the fourth session.
  Arms: Healthy Choices - Motivational Enhancement Intervention
Behavioral: Standard care — Participants will receive standard care plus referrals at three months post-baseline
  Arms: Standard Care

SUMMARY:
Risk behaviors and their associated adverse health outcomes are becoming increasingly problematic among HIV-infected youth. This study is being conducted to test whether a brief motivational enhancement (ME) intervention will help reduce health risk behaviors (drug and alcohol use, sexual risk behavior, poor adherence to medications) among HIV+ youth.

DETAILED DESCRIPTION:
Healthy Choices is a randomized clinical trial examining the efficacy of motivational enhancement in reducing risk and promoting healthy behaviors. This study will use a sample of 225 youth (180 after attrition), ages 16-24, of whom 90 will receive the intervention, referral, and standard care, and 90 will receive referral plus standard care. The sample will be drawn from five study sites. Using parallel screening, recruitment will target 100 youth with an adherence problem, 100 youth with a substance use problem, and 25 youth with a sexual risk problem. A repeated measures design will be used for the proposed study. Primary outcome measures are drug and alcohol use, condom use, and HIV medication adherence. Youth will complete an initial data collection session (baseline) during which questionnaire and interview measures will be administered. Blood specimens for viral load and CD4+ count will also be obtained.

Randomization procedures will take place after completion of the baseline assessment. Participants who are randomized to the intervention group will participate in four sessions for approximately 3 months and will also receive standard care plus individualized referrals. The control group will receive standard care and individualized referrals. All five sites offer comprehensive, multidisciplinary care including social work and case management services and access to mental health services. Participants will receive a three-month post-test designed to coincide with ME completion. Subsequent post-tests will occur at 6, 9, 12, and 15 months after baseline data collection (3, 6, 9, and 12 months after ME completion).

ELIGIBILITY:
Inclusion Criteria:

* HIV infection as documented by professional referral and medical record review. HIV+ participants who are self-referred and not in medical care will be required to provide documentation of test results.
* Males or females between the age of 16 years and 0 days and 24 years and 364 days at the time of study enrollment.
* Reports having ever engaged in at least 2 of the following 3 behaviors based on screening questionnaire:

  * taken prescribed antiretroviral medications, OR been told by his/her physician that he/she should be on antiretroviral medications (whether he/she takes them or not);
  * vaginal or anal sex, OR
  * alcohol or drug use.
* At least one of the 3 aforementioned behaviors are currently at a problem level, based on screening questionnaire:

  * taking currently prescribed antiretroviral medications <90 % of the time in the last month,
  * having unprotected intercourse within the last 3 months,
  * demonstrating problem level alcohol and/or drug use as measured during screening.
* Able to understand spoken and written English sufficiently to provide consent/assent and be interviewed and participate in study intervention.
* Not intending to relocate out of the current geographical area for the duration of study participation.

Exclusion Criteria:

* History of any psychiatric thought disorder (e.g., schizophrenia, schizoaffective disorder).
* Currently involved in behavioral research (assessment or intervention) targeting adherence, sexual risk, or alcohol and/or drug substance abuse OR currently involved in a substance abuse treatment program.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 225 (Actual)
Dates: Start 2005-03; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of a motivational enhancement intervention | 15 months
  The primary objective is to determine the efficacy of a motivational enhancement intervention in reducing health risk behaviors (drug and alcohol use, sexual risk behavior, poor adherence to medications) among HIV+ youth.

SECONDARY OUTCOMES:
Determine the mediators and moderators of the intervention | 15 months
  Determine the mediators (e.g., self-efficacy, stage of change, decisional balance) and moderators (e.g., demographics, emotional distress) of the intervention
Determine secondary intervention effects | 15 months
  Determine secondary intervention effects such as improved health status (through measurements of CD4+ counts and viral load levels), decreased levels of psychological distress, and increased engagement with providers (both medical and ancillary services)
Determine if intervention effects are maintained | 15 months
  Determine if intervention effects are maintained over 12 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Naar-King, PhD, Study Chair — Children's Hospital of Michigan
Locations (6):
- United States (6):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Children's Diagnostic and Teatment Center, Fort Lauderdale, Florida
  - University of Maryland, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naar-King S, Parsons JT, Murphy DA, Chen X, Harris DR, Belzer ME. Improving health outcomes for youth living with the human immunodeficiency virus: a multisite randomized trial of a motivational intervention targeting multiple risk behaviors. Arch Pediatr Adolesc Med. 2009 Dec;163(12):1092-8. doi: 10.1001/archpediatrics.2009.212. PMID 19996045
- See also: description of the Adolescent Trials Network and contact information — http://www.atnonline.org